CLINICAL TRIAL: NCT06347120
Title: Place of Nasogastric Tube in Uncomplicated Adhesive Small Bowel Obstruction : a Randomized Open-label Non-inferiority Trial
Brief Title: Place of Nasogastric Tube in Uncomplicated Adhesive Small Bowel Obstruction
Acronym: BOWNTI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Beauvais (Other); CHU de Rouen - Accueil (Other); Hospital Avicenne (Other); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Limoges (Other); Saint Antoine University Hospital (Other); Centre Hospitalier Universitaire de Besancon (Other); Hôpital Cochin (Other); University Hospital, Toulouse (Other); CH Abbeville (Unknown); University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PI2024_843_0011
Record Dates: First submitted 2024-03-19; First posted 2024-04-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Small Bowel Obstruction Adhesion
Keywords: Small Bowel Obstruction Adhesion; nasogastric tube
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (NGT+ group) (Active Comparator): Patients treated with standard NOM (NGT, intravenous administration of fluids, nill per os, analgesic, antiemetic treatment, and clinical and biochemical monitoring for 72h)
  Interventions: Procedure: nasogastric tube
- Experimental group (NGT- group) (Experimental): Patients treated with NOM without NGT insertion (intravenous administration of fluids, nill per os, analgesic, antiemetic treatment, and clinical and biochemical monitoring for 72h)
  Interventions: Other: NOM without NGT insertion

INTERVENTIONS:
Procedure: nasogastric tube — nasogastric tube (NGT), intravenous administration of fluids, and clinical and biochemical monitoring for 72h.
  Arms: Control group (NGT+ group)
Other: NOM without NGT insertion — intravenous administration of fluids, nill per os, analgesic, antiemetic treatment, and clinical and biochemical monitoring for 72h
  Arms: Experimental group (NGT- group)

SUMMARY:
Acute adhesive Small Bowel Obstruction (ASBO) is a public health issue: this is the 3rd cause of hospitalization in Digestive Surgery Departments, 20-30% of patients will be operated, the mortality rate per episode is 3%, the duration of hospitalization is 8 days (up to 16 if resection), and it is associated with a tremendous health care expenses.

The working group on ASBO of the World Society of Emergency Surgery suggested two distinct approaches for the management of acute ASBO: non-operative management (NOM) which concerning around 85% of patients and operative management (OM) :

* OM: if there is clinical signs of strangulation, peritonitis, bowel ischemia, or if IV CT Scan shows sign of ischemia, strangulation, peritonitis, or if the occlusion persists for more than 72 hours;
* NOM in all other cases, including nasogastric tube (NGT), intravenous administration of fluids, and clinical and biochemical monitoring for 72h.

NGT is an old concept first describe for treatment of ASBO based on several studies made on the dog where he proved efficacy of NGT by aspirating gas in the stomach favorising venous decompression and survival of patients. Since, NGT became one of the pillars of NOM.

However NGT is quite bad tolerated by patients (ranked the most painful hospital procedure), some of them refuse it, others put off after the beginning of the treatment and one of the most frequent complications of NGT is pneumonia, which is quite surprising when the first argument for its insertion is to avoid inhalation pneumonia.

Four specific retrospectives studies showed that absence of NGT is possible in 20 to 80% of included patients and was associated with a decrease: in transit recovery time; in complications rate (including rates of pneumonia); in length of stay (LOS); without an increased risk of surgery or resection. 20-87% (a total of 922 patients) were managed successfully conservatively without NGT with a reduction LOS of 2-6 days compared with NGT. But none of this series focused on the patient relief as an endpoint. A retrospective critical analysis of our own management (January - December 2019, n=96) found that: only 17% of patients had a NGT during the IV CTscan, the presence of the NGT did not influence neither gastric volume nor the rate of full stomach, and gastric volume did not influence patient management.

To summarize, the investigators therefore know that the insertion of a NGT is painful, does not relieve all patients, and has an unquantified therapeutic effect on the evolution of ASBO. That is why it is pertinent, in 2023, to question the useless of NGT in the treatment of ASBO, in selected patients. This study would be the first randomized controlled trial to focus on the absence of NGT for the NOM of patients with ASBO. The results of this study could lead to a change in the surgical practice. The absence of NGT in ASBO management appears to be an innovative practice, in rupture with the current practice. This is a part of the simplification of patients'care suffering from ASBO.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an obstruction believed to be secondary to adhesions (abdominal pain and distention, nausea and/or vomiting, no gas and/or stool).
* Uncomplicated presentation (no signs of strangulation or peritonitis).
* IV CT scan of the abdomen consistent with an uncomplicated ASBO, (performed with a pillow to raise slightly the patient.
* Aged 18 or older.
* Provision of written, informed consent.
* Patient covered by French national health insurance.

Exclusion Criteria:

* An incarcerated and/or strangulated incisional hernia, colonic obstruction.
* No previous abdominal operation.
* Obstruction within 4 weeks after a recent operation.
* Gastrointestinal neoplasm in progress.
* Inflammatory bowel disease in progress.
* Abdominal radiotherapy in the last 6 months.
* Contraindication to intravenous contrast enhancement for the CT scan, pre-existing risks factors for pneumonitis.
* Antecedent of aspiration pneumonia.
* Age > 85 years.
* Orientation disturbance.
* Bedridden.
* Chronic cerebrovascular disease (cerebral infarction sequelae, Parkinson disease etc).
* Dementia.
* Gastroesophageal disorder (gastroesophageal reflux)
* Pregnancy or breastfeeding.
* Patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision).
* Patients unable to provide informed consent.
* Age <18 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Decrease of complication rate in patient without NGT group compared to control group | 3 years
  Decrease of complication rate in patient without NGT group compared to control group

SECONDARY OUTCOMES:
aspiration pneumonia rate in both patient groups | 3 years
  aspiration pneumonia rate in both patient groups

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens Universitary Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No